CLINICAL TRIAL: NCT02434640
Title: Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of BAY1128688 After Multiple Oral Administrations in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 16742; 2014-005298-36 (EudraCT Number)
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — BAY1128688

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BAY1128688 [Dose1] (Experimental): BAY1128688 dose level 1
  Interventions: Drug: BAY1128688
- BAY1128688 [Dose2] (Experimental): BAY1128688 dose level 2
  Interventions: Drug: BAY1128688
- BAY1128688 [Dose3] (Experimental): BAY1128688 dose level 3
  Interventions: Drug: BAY1128688
- BAY1128688 [Dose4] (Experimental): BAY1128688 dose level 4
  Interventions: Drug: BAY1128688
- Placebo (Placebo Comparator): Placebo to match arm 1,2, 3 and 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1128688 — Part A: Single dose and multiple dose for 14 days (postmenopausal women)
  Arms: BAY1128688 [Dose1]; BAY1128688 [Dose2]; BAY1128688 [Dose3]; BAY1128688 [Dose4]
Drug: Placebo — Part A: Single dose and multiple dose for 14 days (postmenopausal women)
  Arms: Placebo
Drug: BAY1128688 — Part B: Multiple dose for 28 days (premenopausal women)
  Arms: BAY1128688 [Dose2]; BAY1128688 [Dose3]

SUMMARY:
The objective of this trial is to investigate the safety and tolerability of BAY1128688 and to determine the concentration of this substance in blood after repeated administration by the oral route. The investigational substance will be administered in tablet form to healthy women.

ELIGIBILITY:
Inclusion Criteria:

PART A

* Postmenopausal state, revealed by

  1. Medical history. One of the following:

     * Natural menopause at least 12 months prior to first study drug administration,
     * Surgical menopause by bilateral ovariectomy at least 3 months prior to first study drug administration) or
     * Hysterectomy AND
  2. Follicle-stimulating hormone (FSH) > 40 IU/L
* Age 45 to 68 years

PART B

* Healthy female subjects

  * Sterilized by tubal-ligation
  * Pre-treatment menstrual cycle assessed as ovulatory
* Completion of more than 3 menstrual cycles after delivery, abortion or lactation
* Age 18 to 48 years

Exclusion Criteria:

* Body mass index (kg/m2) greater or equal 32 (or less or equal 18)
* Smoking: PART A: non-smoking; PART B: less than 10 cigarettes per day
* Use of medicines including but not restricted to contraceptives and NSAIDs (details regarding previous use of medicines provided by the study center)
* Ability and willingness to adhere to restrictions regarding diet (PART A and B) and to eat standardised meals (PART A only)
* Significant diseases of the heart, gastrointestinal tract and/or liver and/or kidney and/or reproductive organs (present or in the past; details will be provided by the study center)
* Recent infectious diseases (details will be provided by the study center)
* Migraine or depression
* Thyroid disease which requires treatment
* Metabolic disorders, for example diabetes mellitus or hypertriglyceridemia
* Drug or alcohol abuse; regular consumption of more than 800 ml of beer per day (or other drinks resembling 40 g of alcohol)

Ages: 18 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Treatment Emergent Adverse Events (TEAEs) with severity grading | Up to 2 months
Cmax,md (maximum concentration) of BAY1128688 after multiple dose | 0, 15, 30, 60, 90min, 2, 3, 4, 6, 8, 12, 24h (24h: QD only)
Cav,md (average steady state concentration) of BAY1128688 after multiple dose | 0, 15, 30, 60, 90min, 2, 3, 4, 6, 8, 12, 24h (24h: QD only)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Neu-Ulm, Bavaria
  - Berlin, State of Berlin

REFERENCES:
- [Derived] Gashaw I, Reif S, Wiesinger H, Kaiser A, Zollmann FS, Scheerans C, Grevel J, Piraino P, Seidel H, Peters M, Rottmann A, Rohde B, Arlt W, Hilpert J. Novel aldo-keto reductase 1C3 inhibitor affects androgen metabolism but not ovarian function in healthy women: a phase 1 study. Eur J Endocrinol. 2023 Jul 10;188(7):578-591. doi: 10.1093/ejendo/lvad063. PMID 37306288